CLINICAL TRIAL: NCT01509742
Title: Effect of NNC 90-1170 on Hypoglycaemic Counterregulation During Stepwise Hypoglycaemic Clamp in Type 2 Diabetic Subjects. A Double-blind, Placebo-controlled, Randomised, 2-period Cross-over Trial
Brief Title: Effect of Liraglutide on Glucagon Secretion in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1224
Record Dates: First submitted 2012-01-06; First posted 2012-01-13 (Estimated); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC 90-1170 (Experimental)
  Interventions: Drug: liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Single dose of 7.5 mcg/kg, injected subcutaneously followed by a hypoglycaemic clamp by concentration measurement
  Other Names: NNC 90-1170
  Arms: NNC 90-1170
Drug: placebo — Single dose injected subcutaneously followed by a hypoglycaemic clamp by concentration measurement
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to examine the effect of NNC 90-1170 on the hypoglycaemic counterregulation in subjects with type 2 diabetes.

ELIGIBILITY:
age: minimum 30, maximum 75 years

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2001-04; Primary Completion 2001-11 (Actual); Study Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
Area under the Curve (AUC) glucagon

SECONDARY OUTCOMES:
Insulin secretion
Glucose
Cortisol
Growth hormone
Adrenaline
Noradrenaline
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bad Lauterberg im Harz, Germany

REFERENCES:
- [Result] Nauck MA, El-Ouaghlidi A, Hompesch M, Jacobsen J, Elbroend B. No Impairment of Hypoglycaemia Counterregulation via Glucagon with the long-acting GLP-1 Derivative, NN2211, in Subjects with Type 2-Diabetes. Diabetologia 2003; 46 (Suppl 2): A285
- [Result] Nauck MA, El-Ouaghlidi A, Hompesch M, Jacobsen J, Elbroend B. No Impairment of Hypoglycemia Counterregulation via Glucagon with NN2211, a GLP-1 Derivative, in Subjects with Type 2-Diabetes. Diabetes 2003; 52 (Suppl 1): A128
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com